CLINICAL TRIAL: NCT05221008
Title: Study on Tolerability, Pharmacokinetics and Pharmacodynamics of SHR6508 in Chinese Patients With Secondary Hyperparathyroidism of Chronic Kidney Disease Treated by Maintenance Hemodialysis
Brief Title: A Trial of SHR6508 in Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR6508-102
Record Dates: First submitted 2022-01-07; First posted 2022-02-02 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Intervention Model Description: SHR6508 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Experimental): Experimental: SHR6508 Placebo Comparator: normal saline
  Interventions: Drug: SHR6508；Placebo
- group B (Experimental): Experimental: SHR6508 Placebo Comparator: normal saline
  Interventions: Drug: SHR6508；Placebo
- group C (Experimental): Experimental: SHR6508 Placebo Comparator: normal saline
  Interventions: Drug: SHR6508；Placebo
- group D (Experimental): Experimental: SHR6508 Placebo Comparator: normal saline
  Interventions: Drug: SHR6508；Placebo

INTERVENTIONS:
Drug: SHR6508；Placebo — Group A:SHR6508 low dose
  Arms: group A
Drug: SHR6508；Placebo — Group B:SHR6508 medium dose
  Arms: group B
Drug: SHR6508；Placebo — Group C:SHR6508 high dose
  Arms: group C
Drug: SHR6508；Placebo — Group D:SHR6508 high dose(single dose)
  Arms: group D

SUMMARY:
The study is being conducted to evaluate the tolerability, pharmacokinetics and pharmacodynamics of SHR6508 for Chinese patients with secondary hyperparathyroidism of chronic kidney disease treated by maintenance hemodialysis

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Diagnosed with end stage renal disease receiving stable hemodialysis
3. Male or female
4. Meet the Body Mass Index standard
5. Conform to the ASA Physical Status Classification
6. Stably use of concomitant medication of other therapies of SHPT
7. Meet the standard of iPTH level, cCa and HB

Exclusion Criteria:

1. Subjects with a history of malignant tumor
2. Subjects with neuropsychiatric diseases
3. Subjects with a history of cardiovascular diseases
4. Subjects with gastrointestinal diseases
5. Subjects with a history of surgery
6. Subjects with a history of blood loss
7. Subjects with a history of parathyroidectomy or planned during the study
8. Subjects with a history of kidney transplant or planned during the study
9. Abnormal blood pressure, serum magnesium, serum transaminase, serum albumin, platelet counts.
10. Subjects with a treatment history of similar drugs
11. Allergic to a drug ingredient or component
12. Pregnant or nursing women
13. No birth control during the specified period of time
14. Subject with a history of alcohol abuse and drug abuse
15. Participated in clinical trials of other drugs (received experimental drugs)
16. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Tmax, Time of maximum observed concentration. | 0 hour to 43 hours after first dose administration
Cmax, Maximum observed concentration. | 0 hour to 43 hours after first dose administration
AUC0-t, Area under the concentration-time curve from time zero to the last measurable concentration. | 0 hour to 43 hours after first dose administration
AUC0-∞, Area under the curve from time 0 extrapolated to infinite time | 0 hour to 43 hours after first dose administration
t1/2z, Terminal elimination half-life | 0 hour to 43 hours after first dose administration
CLz, Total Body Clearance | 0 hour to 43 hours after first dose administration
Vz, Volume of distribution based on the terminal phase | 0 hour to 43 hours after first dose administration
MRT0-t, Mean residence time from time zero to the last measurable concentration. | 0 hour to 43 hours after first dose administration
MRT0-∞, Mean residence time from time 0 extrapolated to infinite time | 0 hour to 43 hours after first dose administration
Cmax,ss : Maximum observed concentration at steady-state. | Day1-Day29(if reach steady-state)
Cmin,ss : Minimum observed concentration at steady-state | Day1-Day29(if reach steady-state)
Cav : Average concentration | Day1-Day29(if reach steady-state)
AUC0-t,ss, Area under the concentration-time curve from time zero to the last measurable concentration at steady-state. | Day1-Day29(if reach steady-state)
AUC0-∞,ss, Area under the concentration-time curve from time 0 extrapolated to infinite time at steady-state. | Day1-Day29(if reach steady-state)
Tmax,ss, Time of maximum observed concentration at steady-state. | Day1-Day29(if reach steady-state)
t1/2z,ss, Terminal elimination half-life at steady-state | Day1-Day29(if reach steady-state)
CLss, Total Body Clearance at steady-state. | Day1-Day29(if reach steady-state)
Vss, Volume of distribution based on the terminal phase at steady-state. | Day1-Day29(if reach steady-state)
MRT0-∞, Mean residence time from time 0 extrapolated to infinite time. | Day1-Day29(if reach steady-state)
DF: Degree of Fluctuation | Day1-Day29(if reach steady-state)
Accumulation Ratio | Day1-Day29(if reach steady-state)

SECONDARY OUTCOMES:
Change From Baseline in serum iPTH, cCa, P, FGF23 and BSAP | 0 hour to 43 hours after first dose administration
  iPTH, FGF23 and BSAP were tested at a central laboratory.
Change From Baseline to End of Study in serum iPTH, cCa, P, FGF23 and BSAP | Day1 to Day29
  iPTH, FGF23 and BSAP were tested at a central laboratory.
Proportion of Participants to End of Study whose iPTH decreased by≥30% from baseline | Day1 to Day29
  iPTH was tested at a central laboratory.
Proportion of Participants to End of Study whose iPTH decreased to 300 pg/mL from baseline | Day1 to Day29
  iPTH was tested at a central laboratory
Participants With Treatment-Emergent Adverse Events (TEAEs) | Day1 to End of Study, End of Study is about Day55
  Terms were coded with Medical Dictionary for Regulatory Activities (MedDRA)

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided